CLINICAL TRIAL: NCT00577538
Title: Prevalence and Risk Factor for Lymphoproliferative Disease in Patients With Inflammatory Bowel Disease
Brief Title: Prevalence of Lymphoma in IBD
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Other Study IDs: 060358; IRB# 0603-58
Record Dates: First submitted 2007-12-19; First posted 2007-12-20 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Lymphoma; Inflammatory Bowel Disease
MeSH Terms: conditions — Lymphoma; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1
- 2

SUMMARY:
Patients with inflammatory bowel disease (IBD) may be at increased risk of lymphoma. The majority of lymphomas in patients with IBD occur in areas of active inflammation. The relationship between IBD and lymphoproliferative disease is however unclear, since both chronic inflammation as well as medications used to treat IBD (especially immunosuppressives - Azathioprine or 6-MP - and anti-TNF alpha agents) have been associated with increased risk of lymphoma. We plan to study the association between IBD and lymphoma in a large, mixed, community based and referral population from the IBD database at Indiana University.

ELIGIBILITY:
Inclusion Criteria:

* Inflammatory Bowel disease
* Lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with both Inflammatory bowel disease and lymphoma over the last 30 years.
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2006-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael V. Chiorean, M.D., Principal Investigator — Indiana University
Locations (1):
- Indiana University Medical Center, Indianapolis, Indiana, United States